CLINICAL TRIAL: NCT05190172
Title: PRO-GLIO: PROton Versus Photon Therapy in IDH-mutated Diffuse Grade II and III GLIOmas
Acronym: PRO-GLIO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Sahlgrenska University Hospital (Other); The Skandion Clinic (Unknown); University Hospital of North Norway (Other); St. Olavs Hospital (Other); Haukeland University Hospital (Other); Lund University Hospital (Other); Ôrebro University Hospital (Unknown); Uppsala University Hospital (Other); Karolinska University Hospital (Other); University Hospital, Umeå (Other); University Hospital, Linkoeping (Other); Jönköping University Hospital (Unknown)
Responsible Party: Principal Investigator, Petter Brandal, Head of Neurooncology, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 265626
Record Dates: First submitted 2021-07-15; First posted 2022-01-13 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Oligodendroglioma; Oligodendroglioma, Anaplastic; Diffuse Astrocytoma, IDH-Mutant
Keywords: proton therapy; radiotherapy; IDH-mutated diffuse grade II astrocytoma; IDH-mutated diffuse grade III astrocytoma; oligodendroglioma
MeSH Terms: conditions — Oligodendroglioma; Astrocytoma | interventions — Radiotherapy

STUDY DESIGN:
Intervention Model Description: * Experimental treatment arm with proton radiationtherapy
  * Standard treatment arm with photon radiationtherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiation therapy with protons (Experimental): Radiation therapy with protons at The Skandion Clinic, Uppsala, Sweden
  Interventions: Radiation: Radiation therapy
- Radiation therapy with photons (Active Comparator): Radiation therapy with photons at an University Hospital nearby subject's home address
  Interventions: Radiation: Radiation therapy

INTERVENTIONS:
Radiation: Radiation therapy — Radiation therapy either with protons or photons

SUMMARY:
Proton therapy is a powerful tool enabling oncologists to spare normal tissue around the target for irradiation much better than what can be achieved with photon irradiation. The infiltrative nature of IDH-mutated grade II and III diffuse glioma, however, renders proton therapy a potential problem. A randomized controlled trial (RCT) is the only option when trying to ensure that chances of long-term survival are not impaired seeking to reduce unwanted late treatment effects. Non-inferiority of proton therapy compared to photon irradiation is the primary endpoint of the RCT.

Hence, PRO-GLIO has two main objectives. First, PRO-GLIO will evaluate if proton therapy is safe in patients with IDH-mutated grade II and III diffuse glioma, showing that survival figures at 2 years from radiotherapy are not poorer in the proton arm than in the photon arm. Second, we want to find the true number of patients in need of rehabilitation in both arms, and evaluate if proton therapy conveys a higher QoL than photon irradiation at 2 years from radiotherapy.

DETAILED DESCRIPTION:
PRO-GLIO aims at establishing proton irradiation as standard radiotherapy for IDH-positive diffuse glioma grade II and III patients. First, PRO-GLIO will show that proton therapy is safe, despite the infiltrative nature of these tumors. Second, the HRQOL and neuropsychological investigating part of PRO-GLIO will show that patients irradiated with protons have a better outcome in this regard than those irradiated with photons. Inclusion criteria are a diagnosis of grade II or grade III IDH-mutated diffuse glioma, good performance status, indication for radiotherapy and age between 18 and 65 years.

Patients will be randomized to proton or photon radiotherapy and the study work will be divided in three work packages (WP).

1. In WP1, survival data will be the main focus, but the estimation of QALY will also be an important part - concentrating on differences between the two study arms. If there is truly no difference between the proton and photon radiotherapy on the probability of FIFS after two years, then 224 randomized patients (112 in each treatment group) are required to be 80% certain that the upper limit of a two-sided 95% confidence interval will exclude a difference in favor of the photon radiotherapy of more than 15%. This assumes a 0.8 probability of FIFS in the control arm, and no drop-outs.
2. In WP2, a battery of validated neuropsychological tests will be used to test the cognive abilities of the patients. All patients will be testes using an internet-based test (Cog-State) and 1/3 of patients will also have an in-depth neuropsychological evaluation. The two methods will be compared.
3. In WP3, a battery of patient-reported outcome measures (PROMS) questionnaires will be used to establish which subjective challenges this patient group struggles the most with.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 18 to 65 years old at the day of consenting
2. IDH-mutated astrocytoma grade II or III, or oligodendroglioma grade II or III according to WHO 2016
3. Indication for radiotherapy
4. WHO/ECOG performance status 0-2
5. Ability to undergo MRI
6. No significant contrast enhancing tumor (more than 1 or 2 punctate contrast enhancing foci) at the time of randomization. In recurrence patients, no contrast enhancement is allowed unless a new biopsy confirms the diagnosis of IDH-mutated astrocytoma grade 2 or 3, or oligodendroglioma grade 2 or 3.
7. Ability and willingness to travel to The Skandion Clinic for proton therapy if randomized to the proton therapy arm
8. Women of child-bearing potential (WOCBP) must agree to use an effective method of contraception during radiotherapy, chemotherapy and 1 year after completion of chemotherapy. Pregnancy is not an ineligibility criterium if radiotherapy is indicated and cannot be postponed
9. Ability to understand the information about the study and included treatment and give a written informed consent
10. Signed informed consent
11. Ability to speak and understand Norwegian or Swedish language

Exclusion Criteria:

1. Prior treatment (except surgery) for diffuse glioma
2. Concomitant or previous malignancies. Exceptions are adequately treated basal cell carcinoma or squamous cell carcinoma of the skin, or in situ carcinoma of the cervix uteri with a follow-up time of at least 3 years, or other previous malignancy with a disease-free interval of at least 5 years
3. Known CDKN2A/B homozygous deletion
4. Presence of any medical, psychological, familial, sociological, or geographical characteristic that might impair patient compliance for study protocol procedures including follow-up
5. Body weight > 150 kg

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Estimated)
Dates: Start 2022-01-14 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2043-12-31 (Estimated)

PRIMARY OUTCOMES:
First intervention free survival (FIFS) at 2 years | 2 years
  Survival

SECONDARY OUTCOMES:
Total fatigue score assessed by the fatigue questionnaire developed by T. Chalder et al. | 2, 5, 10 and 15 years
  Symptom
Change in cognitive functioning (composite score from CANTAB-tests) at 2 years | 5 months and 2, 5, 10 and 15 years
  Objective examination
Overall survival | Median and at 2, 5, 10 and 15 years
  Survival
FIFS | Median, 5, 10 and 15 years
  Survival
Progression-free survival | Median and at 2, 5, 10 and 15 years
  Survival
Change in neurological function as assessed by the NANO scale | 2, 5, 10 and 15 years
  Objective examination
Global cognitive impairment index | 2, 5, 10 and 15 years
  Neuropsychological endpoint
Rate of local, distant and combined recurrences | 2, 5, 10 and 15 years
  Disease development
Rate of patients without epileptic seizures | 5 months and 2, 5, 10 and 15 years
  Symptom
EORTC QLQ C30-based algorithm score | 2, 5, 10 and 15 years
  Quality of life
Incremental cost effectiveness ratio | 2, 5, 10 and 15 years
  Health economics
Rate of adverse events | At 6 weeks, 3 and 5 months and 1 year, 2 , 5, 10 and 15 years
  Toxicity
Costs in Norwegian kroner related to loss of production caused by disease and treatment | 2, 5, 10 and 15 years
  Health economics

CONTACTS AND LOCATIONS:
Overall Officials: Petter Brandal, MD PhD, Principal Investigator — Head of Neurooncology
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Norwegian Data Protection Law, the dataset is only available by physical appearance at Oslo University Hospital, Norway upon request. To access data, please contact principal investigator Petter Brandal (petter.brandal@ous-hf.no). Data will not be shared before planned analyses are performed and published. The study protocol is also available upon request.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available following publication of the primary and key secondary endpoints. The study protocol is available upon request from this date
Access Criteria: Physical appearance at Oslo University Hospital, Norway.

REFERENCES:
- [Derived] Heggebo LC, Borgen IMH, Rylander H, Kiserud C, Nordenmark TH, Hellebust TP, Evensen ME, Gustavsson M, Ramberg C, Sprauten M, Magelssen H, Blakstad H, Moorthy J, Andersson K, Raunert I, Henry T, Moe C, Granlund C, Goplen D, Brekke J, Johannessen TA, Solheim TS, Marienhagen K, Humberset O, Bergstrom P, Agrup M, Dahl L, Gubanski M, Gojon H, Brahme CJ, Ryden I, Jakola AS, Vik-Mo EO, Lie HC, Asphaug L, Hervani M, Kristensen I, Rueegg CS, Olsen IC, Ledal RJ, Degsell E, Werlenius K, Blomstrand M, Brandal P. Investigating survival, quality of life and cognition in PROton versus photon therapy for IDH-mutated diffuse grade 2 and 3 GLIOmas (PRO-GLIO): a randomised controlled trial in Norway and Sweden. BMJ Open. 2023 Mar 20;13(3):e070071. doi: 10.1136/bmjopen-2022-070071. PMID 36940951